CLINICAL TRIAL: NCT07341087
Title: Skin Inflammation in Perimenopause: A Probiotic Intervention Proof of Concept Trial (SIPPI)
Brief Title: Skin Inflammation in Perimenopause: A Probiotic Intervention Proof of Concept Trial
Acronym: SIPPI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Yakult (UK & Ireland) Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HR-25/26-52828; BB/X010821/1 (Other Grant/Funding Number: BBSRC-iNutriLife and Yakult)
Record Dates: First submitted 2025-12-11; First posted 2026-01-14 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-12

CONDITIONS: Acne Vulgaris; Perimenopause; Skin Inflammation; Immunosenescence; Inflammation
Keywords: Perimenopause; Acne vulgaris; Probiotics; Lactobacillus casei Shirota; Immune ageing; Gut-skin axis
MeSH Terms: conditions — Acne Vulgaris; Dermatitis; Inflammation

STUDY DESIGN:
Intervention Model Description: Randomised, parallel, open-label, proof of concept trial, with an 8-week intervention and blinded outcome assessment.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to participant group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 - Probiotic (LcS) (Experimental): Daily 130 ml low-sugar Lactobacillus casei Shirota (LcS) drink for 8 weeks.
  Interventions: Dietary Supplement: Lactobacillus casei Shirota (LcS) Probiotic Drink
- Arm 2 - Control (Active Comparator): Daily 130 ml skimmed milk drink for 8 weeks.
  Interventions: Other: Skimmed Milk Control Drink

INTERVENTIONS:
Dietary Supplement: Lactobacillus casei Shirota (LcS) Probiotic Drink — Daily intake of 130 ml low-sugar fermented milk drink containing Lactobacillus casei Shirota for 8 weeks.
  Arms: Arm 1 - Probiotic (LcS)
Other: Skimmed Milk Control Drink — Daily intake of 130 ml skimmed milk for 8 weeks.
  Arms: Arm 2 - Control

SUMMARY:
This study will explore whether a daily probiotic drink containing Lactobacillus casei Shirota (LcS) can help improve immune function and reduce inflammation in women going through perimenopause. Hormonal changes during this stage of life can affect the immune system, gut health, and skin, sometimes leading to increased inflammation or conditions such as acne.

Participants will consume either a low-sugar LcS probiotic drink or a skimmed milk control drink every day for eight weeks. The study will assess markers of immune ageing, inflammation, skin health, wellbeing, and hormone levels. The results will help determine whether a safe, non-hormonal probiotic approach may support immune and skin health during perimenopause.

DETAILED DESCRIPTION:
Research Question: Can a daily probiotic drink help reduce immune system ageing and improve inflammatory skin conditions, such as acne, in women going through perimenopause?

Background

Perimenopause is the transition before menopause, usually affecting women aged 40-50. During this time, hormone levels, especially oestrogen, fluctuate and gradually decline. These changes can affect the immune system, making it more prone to inflammation and less effective over time.

Lower oestrogen can also affect the skin, leading to dryness, irritation, or acne. It can change the balance of bacteria in the gut and on the skin, which may worsen inflammation and overall health.

While hormone replacement therapy can help some symptoms, it is not suitable for all women. Currently, there is little research on safe, non-hormonal ways to support the gut, immune system, and skin together. One promising approach is using probiotics-beneficial bacteria that can improve gut health and reduce inflammation.

Lactobacillus casei Shirota (LcS) is a probiotic that has shown anti-inflammatory and immune-supporting effects in other adults. However, it has not been studied in perimenopausal women, who are particularly vulnerable to immune system changes and inflammatory skin conditions.

Aims and Hypothesis

Aim: To explore whether an oral probiotic Lactobacillus casei Shirota (LcS) can modulate immunological age markers in perimenopausal women with acne.

Hypothesis: Consuming 130 ml/day of a low-sugar probiotic (LcS) drink for 8 weeks will significantly reduce inflammation in perimenopausal women with acne compared to a 130 ml/day skimmed milk control.

Objectives

Primary Objective: To determine if daily LcS consumption can improve immune function, measured using a composite "immune age" score (IMM-AGE) that reflects overall immune health and inflammation.

Secondary Objectives:

* To look at self-reported skin health, general wellbeing, and gut health.
* To assess skin inflammation and signs of ageing through clinician assessments and images.
* To measure hormone levels (oestrogen and FSH).

Study design

* Trial Design: Randomised, parallel, open-label, proof of concept trial, with an 8-week intervention and blinded outcome assessment.
* Participants: Perimenopausal women aged 40-50 years with self-reported or clinically diagnosed acne.
* Intervention: Daily 130 ml low-sugar LcS probiotic drink for 8 weeks.
* Comparison: Daily 130 ml skimmed milk (control) for 8 weeks.

Measurements:

* Immune function (IMM-AGE)
* Blood markers of inflammation (cytokines including CD14, IFN-α, IFN-γ, IL1Ra, IL-6, IL-10, TNF-α, GM-CSF, IFN-β, IL1β, IL-4, IL-8, IL-17) and hormones (oestrogen and follicle stimulating hormone [FSH] levels)
* Skin health and ageing
* Self-reported wellbeing and gut health

Stool and skin samples will also be collected for future research, but these will not be analysed in this trial.

5. Why This Study Matters

Perimenopause is a time of rapid biological change that can affect immunity and skin health. This trial will test a safe, non-hormonal approach to support the immune system, reduce inflammation, and improve skin health in midlife women. The results will help guide future research and may inform practical strategies to improve wellbeing during perimenopause.

ELIGIBILITY:
Inclusion Criteria:

1. Female, aged 40-50 years, in the perimenopausal transition (defined as menstrual cycle irregularity within the past 12 months but not yet 12 months of amenorrhoea).
2. Clinician-diagnosed acne, defined as the presence of acne symptoms (e.g., comedones, papules, pustules, nodules) or a prior formal diagnosis of acne vulgaris by a healthcare professional.
3. Willing and able to consume a daily oral intervention (2x 65 ml probiotic drinks or skimmed milk) for 8 weeks.
4. Willing and able to provide sufficient blood, skin and stool samples at baseline and end-of-study (Week 8). Participants unable to provide adequate blood sample volumes will not be able to start the intervention.
5. Willing and able to provide a photograph of the facial area, with all images anonymised for study purposes.
6. Able to comply with study procedures, including attending clinic visits at KCL.
7. Have access to a refrigerator at home and be able to store the study product(s) safely after collection (i.e., travel time allows safe storage).
8. Capable of providing written informed consent.
9. Have sufficient proficiency in English to complete study questionnaires and assessments.

Exclusion Criteria:

1. Inability or unwillingness to provide informed consent.
2. Inability or unwillingness to comply with study protocol requirements (e.g., clinic visits, sample provision, daily consumption of study drink)
3. Unwilling to record dietary intakes using handwritten diet diaries
4. Not fluent in the English language
5. Is planning on international travel during the study period
6. Current participation in another interventional clinical trial or having received an investigational/pharmaceutical product within the past 3 months.
7. Known allergy or intolerance to dairy products, skimmed milk, or probiotic drinks containing Lactobacillus species.
8. Currently pregnant, currently breastfeeding or planning to become pregnant in the next 4 months.
9. BMI <18.5kg/m2 or > 35kg/m2.
10. History of substance abuse or alcoholism (alcohol intake >50 units/week) within the last 12 months.
11. Current smokers, or individuals who quit smoking in the last 6-months.
12. Fasting glucose >7mmol/l (finger prick test at baseline clinic).
13. Active skin infection requiring systemic antibiotics, antivirals, or antifungals within the past 4 weeks.
14. Major gastrointestinal disease (e.g., inflammatory bowel disease, celiac disease, short bowel syndrome) or history of significant gastrointestinal surgery (excluding appendectomy or cholecystectomy).
15. Known immunodeficiency (e.g., HIV, immunosuppressive therapy, systemic corticosteroids >10 mg/day prednisolone equivalent).
16. History of malignancy or clinically significant non-malignant skin conditions within the past 5 years (except adequately treated basal cell carcinoma).
17. Serious medical conditions that, in the opinion of the investigator, would compromise safety or interfere with study outcomes (e.g., uncontrolled diabetes, advanced cardiovascular, hepatic, or renal disease, active cancer).
18. Women with a history of severe psychiatric illness that would limit adherence to study requirements.
19. Current use of probiotics, prebiotics, or antibiotics within 4 weeks prior to baseline.
20. Current use of systemic corticosteroids, or other immunosuppressive/immunomodulatory therapies within the past 3 months.
21. Currently receiving, or having received, phototherapy (e.g., UVB, PUVA, laser/light-based treatments, including at home treatments) for any skin condition within the past 3 months.
22. Currently receiving, or having received, systemic dermatology treatments likely to affect skin inflammation or immune response within the past 3 months (e.g., isotretinoin, methotrexate, cyclosporine, biologics such as TNF, IL-17, IL-23 or IL-4/IL-13 inhibitors).
23. Currently receiving, or having received, topical treatments likely to significantly alter skin inflammation within the past 3 months (e.g., high-potency topical corticosteroids, topical calcineurin inhibitors such as tacrolimus or pimecrolimus, topical retinoids, or photodynamic therapy).
24. Currently using, or have used, probiotic skincare (e.g., topical creams and serums) within the past 3 months.
25. Currently receiving, have undergone, or plan to undergo cosmetic skin procedures (e.g., chemical peels, laser therapy, dermal fillers, microneedling) within the 3 months prior to, or within 3 months after the first (baseline) visit.
26. Currently using, or have used, hormonal contraceptives or treatments known to exacerbate acne, including Mirena (levonorgestrel-releasing intrauterine system), oral progesterone-only contraceptives (e.g., mini-pill), and synthetic progestogens (e.g., norethisterone) within the past 3 months.
27. Habitual dietary fibre intake below 10g/day, assessed via the screening questionnaire or dietary assessment, due to the potential impact of low fibre intake on the gut microbiome and study outcomes.

Ages: 40 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03-09 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Immunological age (IMM-AGE) composite scores | Baseline (Week 0) and end of intervention (Week 8).
  A subset of eight immune cell types-total T cells, naïve CD4 T cells, effector memory CD4 T cells, effector memory CD8 T cells, EMRA CD8 T cells, CD28- CD8 T cells, CD57⁺ CD8 T cells, and regulatory T cells-will be used to generate a composite score ranging from 0 to 1 that reflects the degree of immune ageing. Higher scores indicate more advanced immune ageing and worse outcomes.
Serum inflammaging markers | Baseline (Week 0) and end of intervention (Week 8).
  Serum cytokines including CD14, IFN-α, IFN-γ, IL-1Ra, IL-6, IL-10, TNF-α, GM-CSF, IFN-β, IL-1β, IL-4, IL-8, and IL-17.

SECONDARY OUTCOMES:
Acne-related quality of life | Baseline (Week 0), Midpoint (Week 4) and Endpoint (Week 8)
  Health-related quality of life will be assessed using the Dermatology Life Quality Index (DLQI), a validated, self-administered questionnaire for individuals with skin conditions such as acne. The DLQI consists of 10 items, each scored from 0 ("Not at all" or "Not relevant") to 3 ("Very much"). Total scores range from 0 to 30, where 0 represents no impact on quality of life and 30 represents an extremely large negative impact. Higher scores indicate worse health-related quality of life outcomes.
Acne severity - participant perception | Baseline (Week 0), Midpoint (Week 4) and Endpoint (Week 8)
  The Patient Global Assessment (PtGA) will be used to assess the participant's overall perception of their acne severity. The PtGA is a patient-reported outcome measure scored on a numeric scale ranging from 0 to 10, where 0 represents no symptoms and 10 represents the worst possible acne symptom severity imaginable. Higher scores indicate worse acne severity and worse outcomes.
Acne severity - clinician rated (measure 1) | Baseline (Week 0), Midpoint (Week 4) and Endpoint (Week 8)
  Acne severity will be assessed by a blinded clinician using standardised photographic images and the Leeds Acne Grading System, with scores ranging from 0 to 10. Higher scores indicate more severe acne and worse outcomes.
Acne severity - clinician rated (measure 2) | Baseline (Week 0), Midpoint (Week 4) and Endpoint (Week 8)
  Acne severity will be assessed by a blinded clinician using standardised photographic images and the Investigator Global Assessment (IGA), scored from 0 (clear) to 4 (severe). Higher scores indicate worse outcomes.
Skin Ageing | Baseline (Week 0), Midpoint (Week 4) and Endpoint (Week 8)
  Signs of skin ageing will be assessed by a blinded clinician using standardised photographic images and the Griffiths Photonumeric Scale. The Griffiths scale is a validated 9-point photonumeric grading system used to assess the severity of facial photoaging features, including wrinkling, pigmentation changes, and overall skin texture. Scores range from 0 (no photoaging) to 8 (severe photoaging), with higher scores indicating more advanced skin ageing and worse outcomes.
General wellbeing | Baseline (Week 0) and Endpoint (Week 8)
  Wellbeing will be assessed using the World Health Organization Five Well-Being Index (WHO-5), a validated, self-administered questionnaire measuring current mental wellbeing. The WHO-5 consists of five items, each scored from 0 ("At no time") to 5 ("All of the time"). Raw total scores range from 0 to 25, with higher scores indicating better wellbeing. For standardised reporting, the total score may be transformed to a scale from 0 to 100, where 0 represents the worst possible wellbeing and 100 represents the best possible wellbeing.
Menopause symptoms | Baseline (Week 0), Midpoint (Week 4) and Endpoint (Week 8)
  Menopausal symptoms will be assessed using the Menoscale, a questionnaire consisting of 20 questions about menopausal symptoms. For each symptom, participants rate the extent to which it impacts their life using a scale from 0 ("Not at all") to 5 ("Extremely"). Responses are summed to generate a total score ranging from 0 to 100. Higher scores indicate a greater burden of menopausal symptoms and a worse impact on quality of life.
Anxiety symptoms | Baseline (Week 0), Midpoint (Week 4) and Endpoint (Week 8)
  Anxiety symptoms will be assessed using the Generalized Anxiety Disorder 7-item scale (GAD-7), a validated, self-administered questionnaire. The GAD-7 consists of seven items, each scored from 0 ("Not at all") to 3 ("Nearly every day"). Total scores range from 0 to 21, with higher scores indicating more severe anxiety symptoms and worse outcomes.
Depressive symptoms | Baseline (Week 0), Midpoint (Week 4) and Endpoint (Week 8)
  Depressive symptoms will be assessed using the Patient Health Questionnaire-9 (PHQ-9), a validated, self-administered questionnaire. The PHQ-9 consists of nine items, each scored from 0 ("Not at all") to 3 ("Nearly every day"). Total scores range from 0 to 27, with higher scores indicating more severe depressive symptoms and worse outcomes.
Gastrointestinal symptoms | Baseline (Week 0), Midpoint (Week 4) and Endpoint (Week 8)
  Gastrointestinal symptoms will be assessed using the Gastrointestinal Symptom Rating Scale (GSRS), a validated, self-administered questionnaire. The GSRS consists of multiple items assessing gastrointestinal symptoms, each scored on a Likert scale from 1 to 7. Item scores are averaged to generate a total score ranging from 1 to 7, where 1 represents no discomfort and 7 represents very severe discomfort. Higher scores indicate worse gastrointestinal symptom severity and worse outcomes.
Stool consistency | Baseline (Week 0) and Endpoint (Week 8)
  Stool form will be assessed using the Bristol Stool Form Scale (BSFS), a validated visual and descriptive scale used to classify stool consistency. The BSFS categorises stool form into seven types, ranging from Type 1 (separate hard lumps, indicating severe constipation) to Type 7 (watery, no solid pieces, indicating severe diarrhoea). Lower scores indicate harder stool consistency, and higher scores indicate looser stool consistency and worse gastrointestinal outcomes.
Body weight | Baseline (Week 0), Midpoint (Week 4) and Endpoint (Week 8)
  Body weight will be measured in kilograms (kg) using a calibrated scale. Changes in body weight will be assessed over time, with higher values indicating greater body weight.
Body Mass Index (BMI) | Baseline (Week 0), Midpoint (Week 4), Endpoint (Week 8)
  Body mass index (BMI) will be calculated as weight in kilograms divided by height in meters squared (kg/m²). Higher BMI values indicate greater body mass relative to height.
Body fat percentage | Baseline (Week 0), Midpoint (Week 4), Endpoint (Week 8)
  Body fat percentage will be measured using a bioelectrical impedance analysis (BIA) scale and reported as a percentage (%). Higher values indicate a greater proportion of body fat.
Waist circumference | Baseline (Week 0), Midpoint (Week 4), Endpoint (Week 8)
  Waist circumference will be measured in centimetres (cm) using a standardised tape measure at the midpoint between the lowest rib and the iliac crest. Higher values indicate greater central adiposity.
Hip circumference | Baseline (Week 0), Midpoint (Week 4), Endpoint (Week 8)
  Hip circumference will be measured in centimetres (cm) using a standardised tape measure at the level of the widest portion of the buttocks. Higher values indicate greater hip circumference.
Systolic Blood Pressure | Baseline (Week 0), Midpoint (Week 4), Endpoint (Week 8)
  Systolic blood pressure will be measured in millimetres of mercury (mmHg) using a calibrated sphygmomanometer. Higher values indicate higher systolic blood pressure and worse cardiovascular outcomes.
Diastolic blood pressure | Baseline (Week 0), Midpoint (Week 4), Endpoint (Week 8)
  Diastolic blood pressure will be measured in millimetres of mercury (mmHg) using a calibrated sphygmomanometer. Higher values indicate higher diastolic blood pressure and worse cardiovascular outcomes.

OTHER OUTCOMES:
Hormone levels | Baseline (Week 0)
  Follicle Stimulating Hormone (FSH) and oestrogen levels - to control for heterogeneity in peri-menopausal status
Ovarian reserve | Baseline (Week 0)
  The Stages of Reproductive Aging Workshop +10 (STRAW+10) criteria will be used to classify reproductive aging stage and to determine ovarian reserve and perimenopausal status based on menstrual cycle characteristics and relevant clinical information. Classification will be performed according to established STRAW+10 definitions.
Fasting glucose levels | Baseline (Week 0)
  Fasting blood glucose levels will be measured using a finger-prick capillary blood test after an overnight fast. This will be used to screen for (and exclude those with) hyperglycaemia (>7 mmol/L).

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Hall, Principal Investigator — King's College London; Andrea Du Preez, Study Director — King's College London
Locations (1):
- Metabolic Research Unit, 4th Floor (Corridor A), Franklin-Wilkins Building, KCL., London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared outside the study team because our ethics approval and participant consent do not permit external sharing of de-identified data.